CLINICAL TRIAL: NCT07249138
Title: Impact of Congenital Heart Disease on Quality of Life and Long-Term Outcomes in Childhood Hematological Tumor Survivors
Brief Title: Impact of Congenital Heart Disease on the Prognosis of Childhood Hematological Neoplasms: A Multicenter Cohort Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Nanjing Children's Hospital (Other); Children's Hospital of Suzhou University (Unknown); Tongji Hospital (Other); Shandong Provincial Hospital (Other Government); Guangzhou Women and Children's Medical Center (Other); Wuhan Children's Hospital (Other); Union Hospital of Huazhong University of Science and Technology (Unknown); The Third Xiangya Hospital of Central South University (Other); Inner Mongolia Maternal and Child Health Care Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Beijing Children's Hospital (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Shanxi Provincial Maternity and Children's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Shanghai Children's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHOPA0012-CHFUCHD-2023
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Disease (CHD); Hematologic Malignancy
MeSH Terms: conditions — Heart Defects, Congenital; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow Mononuclear Cells (BMMCs) in TRIzol (-80°C) Serum and Plasma aliquots (-80°C) Peripheral Blood Mononuclear Cells (PBMCs) (-80°C or in liquid nitrogen) Genomic DNA from blood or bone marrow (-80°C) Genomic RNA from blood or bone marrow (-80°C)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort of pediatric patients with congenital heart disease and hematological tumors
- Cohort of pediatric patients with hematological tumors

SUMMARY:
This study aims to determine whether congenital heart disease increases chronic health risks and mortality in childhood hematological tumor survivors, explore potential shared genetic factors between these conditions, identify other factors affecting long-term outcomes and quality of life, and validate any discovered genetic links through mechanistic investigations.

DETAILED DESCRIPTION:
Children with congenital heart disease have a significantly higher risk of developing hematological tumors compared to the general pediatric population, although the clinical characteristics and prognosis of such comorbid cases have previously lacked systematic investigation. The study is set to include children with comorbid congenital heart disease and hematological tumors, comparing them with those without congenital heart disease, to conduct a detailed analysis of their clinical data, treatment responses, and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Children with hematologic malignancies diagnosed by pathology or bone marrow aspiration/biopsy at member hospitals of the Hematologic Oncology Specialty Alliance between 2010 and 2025;
2. Aged 0-17 years at diagnosis, regardless of gender;
3. Completed standard treatment for hematologic malignancies and confirmed diagnosis of congenital heart disease by cardiac ultrasound and clinical evaluation;
4. Written informed consent can be provided by the child or their legal guardian.

Exclusion Criteria:

1. Presence of birth defects other than congenital heart disease;
2. Other serious cardiac conditions, malignancies, or comorbidities that may interfere with study results;
3. Inability to provide the information and data required for the study.

Ages: 0 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will comprise pediatric patients with hematological malignancies who also have congenital heart disease, identified through a multi-center collaborative network spanning major tertiary hospitals across China. This cohort will include children aged 0-18 years at diagnosis who were treated between 2010 and 2025, with detailed clinical data collected retrospectively from participating medical institutions. The selection specifically focuses on patients who completed standard oncologic treatment and received confirmed congenital heart disease diagnoses through comprehensive cardiac evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of all-cause death | from enrollment to follow-up for 5 year
Frequency and severity of SAEs assessed by CTCAE v5.0 | from enrollment to follow-up for 5 year
  CommonTerminology Criteria for Adverse Events（CTCAE）has 5 levels of AE determination, increasing in severity as the level increases

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Children's Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - Guangzhou Women and Children's Medical Center, Guangzhou
  - Inner Mongolia Maternal and Child Health Care Hospital, Hohhot
  - Shandong Provincial Hospital, Jinan
  - Nanjing Children's Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's HospitalShanghai Children's Hospital, Shanghai
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Children's Hospital of Soochow University, Suzhou
  - Shanxi Children's Hospital, Taiyuan
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan
  - Union Hospital of Huazhong University of Science and Technology, Wuhan
  - Wuhan Children's Hospital, Wuhan
  - Northwest Women's and Children's Hospital, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou